CLINICAL TRIAL: NCT04437940
Title: Evaluation of Vaginal Fluid for Covid-19 Positivity
Brief Title: Evaluation of Vaginal Fluid for Covid-19 Positivity in Women With Positive Nasofarengeal Covid-19 Test
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Ozguc Takmaz, MD,Assistant Professor, Acibadem University
Other Study IDs: Acibadem Maslak Ob&Gyn
Record Dates: First submitted 2020-06-17; First posted 2020-06-18 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: COVID; Sars-CoV2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vaginal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid-19 positive women: Women with nasofarangeal Covid-19 PCR test is positive
  Interventions: Diagnostic Test: Vaginal fluid Covid-19 PCR test

INTERVENTIONS:
Diagnostic Test: Vaginal fluid Covid-19 PCR test — Vaginal fluid samples are tested for Covid-19

SUMMARY:
Aim of the study is to investigate whether the Covid-19 is found in the vaginal swab samples of female patients diagnosed with covid-19, to evaluate the presence of Covid-19 and the risk of transmission of Covid-19 by intercourse or vaginal delivery.

DETAILED DESCRIPTION:
Vaginal Covid-19 will be tested by taking vaginal swabs from female patients whose clinical findings are compatible with Covid-19 in Acıbadem Maslak Hospital. In patients with positive vaginal Covid-19 test, vaginal Covid-19 will be re-evaluated for the assessment of viral clearance.

ELIGIBILITY:
Inclusion Criteria:

* Women who are positive nasofarengeal Covid-19 PCR test result
* Women who are 18 years or older
* Women who had sexual intercourse before

Exclusion Criteria:

* who had medical treatment for Covid-19

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who are older than 18 years old Women who had sexual intercourse before
Study Population: Women who are older than18 years old, who are considered to be covid-19 clinically and radiologically positive or nasofarengeal Covid-19 PCR test is positive will be included.
  Patients previously treated for covid-19 will be excluded from the study.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Vaginal fluid Covid-19 PCR test result | 1 month
  Vaginal fluid Covid-19 test positivity rate for patients whose nasofarengeal test is positive

SECONDARY OUTCOMES:
becoming negative from positive | 2 month
  The ratio of negative test results to previous positive results for vaginal fluid Covid-19 test

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem Maslak Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data of the patients will be shared without personel informations

REFERENCES:
- [Background] Cui P, Chen Z, Wang T, Dai J, Zhang J, Ding T, Jiang J, Liu J, Zhang C, Shan W, Wang S, Rong Y, Chang J, Miao X, Ma X, Wang S. Severe acute respiratory syndrome coronavirus 2 detection in the female lower genital tract. Am J Obstet Gynecol. 2020 Jul;223(1):131-134. doi: 10.1016/j.ajog.2020.04.038. Epub 2020 May 4. No abstract available. PMID 32376320
- [Result] Qiu L, Liu X, Xiao M, Xie J, Cao W, Liu Z, Morse A, Xie Y, Li T, Zhu L. SARS-CoV-2 Is Not Detectable in the Vaginal Fluid of Women With Severe COVID-19 Infection. Clin Infect Dis. 2020 Jul 28;71(15):813-817. doi: 10.1093/cid/ciaa375. PMID 32241022